CLINICAL TRIAL: NCT02603393
Title: A 26-week, Randomized, Double Blind, Parallel-group Multicenter Study to Assess the Efficacy and Safety of QVA149 (110/50 μg o.d.) vs Tiotropium (18 µg o.d.) + Salmeterol/Fluticasone Propionate FDC (50/500 µg b.i.d.) in Patients With Moderate to Severe COPD
Brief Title: Evaluation of the Efficacy and Safety of QVA149 (110/50 μg o.d.) vs Tiotropium (18 µg o.d.) + Salmeterol/Fluticasone Propionate FDC (50/500 µg b.i.d.) in Patients With Moderate to Severe COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQVA149A2316; 2015-000114-22 (EudraCT Number)
Record Dates: First submitted 2015-09-17; First posted 2015-11-11 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD, QVA149
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol-glycopyrronium combination; Tiotropium Bromide; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- QVA149 (Experimental)
  Interventions: Drug: QVA149
- Tiotropium + salmeterol/fluticasone (Active Comparator)
  Interventions: Drug: Tiotropium; Drug: Salmeterol/fluticasone

INTERVENTIONS:
Drug: QVA149 — QVA149 will be supplied in a capsule form in blister packs for use in the Novartis Concept 1 SDDPI
  Arms: QVA149
Drug: Tiotropium — Tiotropium will be supplied as commercially available blisters, delivered via HandiHaler®
  Arms: Tiotropium + salmeterol/fluticasone
Drug: Salmeterol/fluticasone — Salmeterol/fluticasone propionate dry inhalation powder delivered via Accuhaler™
  Arms: Tiotropium + salmeterol/fluticasone

SUMMARY:
This study will evaluate the efficacy and safety of QVA149 (110/50 μg o.d.) vs tiotropium (18 µg o.d.) + salmeterol/fluticasone propionate FDC (50/500 µg b.i.d.) in patients with moderate to severe COPD

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed Informed Consent Form prior to initiation of any study-related procedure.
* Male and female adults aged ≥ 40 years.
* Patients with moderate to severe airflow obstruction with stable COPD (Stage 2 or Stage 3) according to the 2014 GOLD Guidelines.
* Patients with a post-bronchodilator FEV1 ≥40 and < 80% of the predicted normal value, and post-bronchodilator FEV1/FVC < 0.70 at run-in Visit 101. (Post refers to 15 min after inhalation of 400 µg of salbutamol).
* Current or ex-smokers who have a smoking history of at least 10 pack years (e.g. 10 pack years = 1 pack /day x 10 years, or ½ pack/day x 20 years). An ex-smoker is defined as a patient who has not smoked for ≥ 6 months at screening.
* Patients who are on triple treatment at least for the last 6 months (LAMA +LABA/ICS).

Exclusion Criteria:

* Patients who have not achieved acceptable spirometry results at Visit 101 in accordance with ATS (American Thoracic Society)/ERS (European Respiratory Society) criteria for acceptability (one retest may be performed for patients that don't meet the acceptability criteria) .
* Patients who have had more than one COPD exacerbation that required treatment with antibiotics and/or oral corticosteroids and/or hospitalization in the last year prior to Visit 1.
* Patients who developed a COPD exacerbation of any severity either 6 weeks before the screening (Visit 1) or between screening (Visit 1) and treatment (Visit 201) will not be eligible but will be permitted to be re-screened after a minimum of 6 weeks after the resolution of the COPD exacerbation.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2017-07-18 (Actual); Study Completion 2017-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (136):
- Argentina (9):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Lanús, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, Concepción del Uruguay, Entre Ríos Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Ciudad Autonoma de Bs As
  - Novartis Investigative Site, Mendoza
- Austria (5):
  - Novartis Investigative Site, Amstetten
  - Novartis Investigative Site, Feldbach
  - Novartis Investigative Site, Feldkirch
  - Novartis Investigative Site, Grieskirchen
  - Novartis Investigative Site, Thalheim bei Wels
- Belgium (5):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Erpent
  - Novartis Investigative Site, Éghezée
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Turnhout
- Bulgaria (4):
  - Novartis Investigative Site, Gabrovo
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Stara Zagora
  - Novartis Investigative Site, Varna
- Canada (8):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Burlington, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Gatineau, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Saint-Charles-Borromée, Quebec
  - Novartis Investigative Site, Victoriaville, Quebec
- Croatia (2):
  - Novartis Investigative Site, Rijeka, HRV
  - Novartis Investigative Site, Zagreb
- Czechia (5):
  - Novartis Investigative Site, Mělník, Czech Republic
  - Novartis Investigative Site, Benešov
  - Novartis Investigative Site, Brandýs nad Labem
  - Novartis Investigative Site, Kyjov
  - Novartis Investigative Site, Pilsen
- Denmark (2):
  - Novartis Investigative Site, Copenhagen NV
  - Novartis Investigative Site, Hvidovre
- Estonia (3):
  - Novartis Investigative Site, Kohtla-Järve
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Germany (26):
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Peine, Lower Saxony
  - Novartis Investigative Site, Warendorf, North Rhine-Westphalia
  - Novartis Investigative Site, Koblenz, Rhineland-Palatinate
  - Novartis Investigative Site, Cottbus, Saxony
  - Novartis Investigative Site, Bad Wörishofen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Menden
  - Novartis Investigative Site, Neu-Isenburg
  - Novartis Investigative Site, Oschatz
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Schleswig
  - Novartis Investigative Site, Solingen
  - Novartis Investigative Site, Wiesloch
- Greece (3):
  - Novartis Investigative Site, Heraklion - Crete, Greece
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
- Hungary (5):
  - Novartis Investigative Site, Százhalombatta, HUN
  - Novartis Investigative Site, Törökbálint, Pest County
  - Novartis Investigative Site, Balassagyarmat
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szekszárd
- Latvia (7):
  - Novartis Investigative Site, Balvi, LVA
  - Novartis Investigative Site, Jūrmala, LVA
  - Novartis Investigative Site, Liepāja, LV
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Krāslava
  - Novartis Investigative Site, Riga
- Lithuania (4):
  - Novartis Investigative Site, Kaunas, LT
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Utena
  - Novartis Investigative Site, Vilnius
- Netherlands (4):
  - Novartis Investigative Site, Alkmaar
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Zutphen
- Poland (12):
  - Novartis Investigative Site, Wroclaw, Lower Silesian Voivodeship
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Bieńkówka
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Ostrów Wielkopolski
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Sopot
  - Novartis Investigative Site, Tarnów
  - Novartis Investigative Site, Wroclaw
  - Novartis Investigative Site, Ostrowiec Swietokrzyskie, Świętokrzyskie Voivodeship
- Romania (7):
  - Novartis Investigative Site, Bucharest, District 1
  - Novartis Investigative Site, Timișoara, Timiș County
  - Novartis Investigative Site, Arad
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Deva
- Serbia (5):
  - Novartis Investigative Site, Belgrade, Serbia
  - Novartis Investigative Site, Belgrade
  - Novartis Investigative Site, Knez-Selo
  - Novartis Investigative Site, Kragujevac
  - Novartis Investigative Site, Valjevo
- Slovakia (4):
  - Novartis Investigative Site, Humenné
  - Novartis Investigative Site, Poprad
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Spišská Nová Ves
- Spain (8):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Centelles, Barcelona
  - Novartis Investigative Site, Ponferrada, Castille and León
  - Novartis Investigative Site, Canet de Mar, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Mérida, Extremadura
  - Novartis Investigative Site, Alzira, Valencia
  - Novartis Investigative Site, Sant Joan d'Alacant, Valencia
- United Kingdom (8):
  - Novartis Investigative Site, Royal Leamington Spa, Warwickshire
  - Novartis Investigative Site, Crawley, West Sussex
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Bath
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Coventry
  - Novartis Investigative Site, Plymouth
  - Novartis Investigative Site, Wolverhampton

REFERENCES:
- [Derived] Chapman KR, Hurst JR, Frent SM, Larbig M, Fogel R, Guerin T, Banerji D, Patalano F, Goyal P, Pfister P, Kostikas K, Wedzicha JA. Long-Term Triple Therapy De-escalation to Indacaterol/Glycopyrronium in Patients with Chronic Obstructive Pulmonary Disease (SUNSET): A Randomized, Double-Blind, Triple-Dummy Clinical Trial. Am J Respir Crit Care Med. 2018 Aug 1;198(3):329-339. doi: 10.1164/rccm.201803-0405OC. PMID 29779416

RESULTS

PARTICIPANT FLOW:
Groups:
- QVA149: 110/50 μg capsules o.d. for inhalation
- Tiotropium + Salmeterol/Fluticasone: tiotropium (18 μg o.d.), and salmeterol/fluticasone propionate FDC (50/500 μg b.i.d.)
Period: Overall Study
Arm/Group | QVA149 | Tiotropium + Salmeterol/Fluticasone
Started | 527 | 526
Completed | 456 | 472
Not Completed | 71 | 54
Not completed — Patient/guardian decision | 32 | 18
Not completed — Adverse Event | 17 | 15
Not completed — Technical problems | 4 | 7
Not completed — Lack of Efficacy | 7 | 2
Not completed — Death | 3 | 4
Not completed — Physician Decision | 3 | 3
Not completed — Protocol deviation | 2 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Non-compliance with study treatment | 1 | 0
Not completed — Sponsor decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QVA149 | Tiotropium + Salmeterol/Fluticasone | Total
Number analyzed (Participants) | 527 | 526 | 1053
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (7.99) | 65.2 (7.62) | 65.3 (7.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 161 | 310
  Male | 378 | 365 | 743
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 526 | 523 | 1049
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Post-dose Trough FEV1
Description: Mean change from baseline in post-dose trough forced expiratory volume in 1 second (FEV1) following 26 weeks of treatment. Trough FEV1 is defined as the mean of the two FEV1 values measured at 23 hr 15 min and 23 hr 45 min after the morning dose taken at site on Day 181. Baseline FEV1 is defined as the average of the pre-dose FEV1 measured at -45 min and -15 min at Day 1.
Time Frame: Baseline, 26 weeks
Population: Full Analysis Set: The full analysis set included all randomized participants who received at least one dose of study drug. Patients in the FAS were analyzed according to the treatment they were randomized to.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Tiotropium + Salmeterol/Fluticasone
Number analyzed (Participants) | 527 | 526
Liters | -0.029 (0.0119) | -0.003 (0.0115)
Statistical Analysis 1: Comparison: QVA149 vs Tiotropium + Salmeterol/Fluticasone; Test type: Non-Inferiority — Non-inferiority will be demonstrated if the 95% confidence interval of the treatment difference lies entirely to the right of (higher than) -50 mL; p = 0.0404, Mixed Model for Repeated Measures Analys — 1 sided; Mean Difference (Final Values) = -0.026, 95% CI [-0.053 to 0.001]

2. Secondary Outcome: Annualized Rate of Moderate or Severe COPD Exacerbations
Description: Moderate or severe COPD exacerbations starting between first dose and one day after last treatment are included. COPD exacerbations that occurred within 7 days of each other are collapsed as one event.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: COPD exacerbations/year
Arm/Group | QVA149 | Tiotropium + Salmeterol/Fluticasone
Number analyzed (Participants) | 527 | 526
COPD exacerbations/year | 0.52 [0.43 to 0.63] | 0.48 [0.40 to 0.58]
Statistical Analysis 1: Comparison: QVA149 vs Tiotropium + Salmeterol/Fluticasone; Test type: Superiority; p = 0.5802, Generalized Linear Model Analysis — 2 sided; Ratio of rates = 1.08, 95% CI [0.83 to 1.40]

3. Secondary Outcome: Annualized Rate of COPD Exacerbations Requiring Treatment With Systemic Glucocorticosteroids and/or Antibiotics, Moderate Exacerbations Only
Description: COPD exacerbations starting between first dose and one day after last treatment are included. COPD exacerbations that occurred within 7 days of each other are collapsed as one event
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: COPD Exacerbations/year
Arm/Group | QVA149 | Tiotropium + Salmeterol/Fluticasone
Number analyzed (Participants) | 527 | 526
COPD Exacerbations/year | 0.47 [0.39 to 0.58] | 0.44 [0.36 to 0.53]
Statistical Analysis 1: Comparison: QVA149 vs Tiotropium + Salmeterol/Fluticasone; Test type: Superiority; p = 0.5651, Generalized Linear Model Analysis — 2-sided; Ratio of rates = 1.08, 95% CI 2-sided [0.82 to 1.43]

4. Secondary Outcome: Annualized Rate of COPD Exacerbations Requiring Hospitalisation
Description: as for outcome 3
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: COPD Exacerbations/year
Arm/Group | QVA149 | Tiotropium + Salmeterol/Fluticasone
Number analyzed (Participants) | 527 | 526
COPD Exacerbations/year | 0.001 [0.0 to NA] — NA - Not estimable No patient in either treatment group had an event | 0.001 [0.00 to NA] — NA - Not estimable No patient in either treatment group had an event
Statistical Analysis 1: Comparison: QVA149 vs Tiotropium + Salmeterol/Fluticasone; Test type: Superiority; p = 0.9665, Generalized Linear Model Analysis — 2-sided; Ratio of rates = 1.02, 95% CI 2-sided [0.44 to 2.34]

5. Secondary Outcome: Mean Change From Baseline in Pre-dose Trough FEV1
Description: Trough FEV1 is defined as the average of the pre-dose FEV1 measurements at -45 min and -15 min prior to dosing at each visit except Day 182 which is the average of the post-dose FEV1 measurements at 23h15min and 23h45min after dosing at Day 181. Baseline FEV1 is considered the Day 1 average of pre-dose measurements.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Tiotropium + Salmeterol/Fluticasone
Number analyzed (Participants) | 527 | 526
Liters | -0.029 (0.0119) | -0.003 (0.0115)
Statistical Analysis 1: Comparison: QVA149 vs Tiotropium + Salmeterol/Fluticasone; Test type: Superiority; p = 0.0573, Mixed Model for Repeated Measures Analys — 2-Sided; Mean Difference (Final Values) = -0.026, 95% CI [-0.053 to 0.001]

6. Secondary Outcome: Mean Change From Baseline in St. George's Respiratory Questionnaire
Description: The St. George Respiratory Questionnaire C (SGRQ-C) is used to provide the health status measurements in this study. Baseline SGRQ-C is defined as the assessment taken right before the first dose of the double-blind drug on Day 1. Higher values correspond to greater impairment of health status. The SGRQ contains 50 items divided into 2 parts covering 3 aspects of health related to COPD: Part I covers "Symptoms" and is concerned with respiratory symptoms, their frequency and severity; Part II covers "Activity" and is concerned with activities that cause or are limited by breathlessness; Part II is also concerned with "Impacts", which covers a range of aspects concerned with social functioning and psychological disturbances resulting from airways disease. A score was calculated for each of these 3 subscales and a "Total" score was calculated. In each case the lowest possible value is zero and the highest 100. Higher values correspond to greater impairment of health status.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QVA149 | Tiotropium + Salmeterol/Fluticasone
Number analyzed (Participants) | 527 | 526
Score on a scale | -0.7 (0.53) | -2.5 (0.51)
Statistical Analysis 1: Comparison: QVA149 vs Tiotropium + Salmeterol/Fluticasone; Test type: Superiority; p = 0.0022, Mixed Model for Repeated Measures Analys — 2-Sided; Mean Difference (Final Values) = 1.8, 95% CI [0.7 to 3.0]

7. Secondary Outcome: Mean Change From Baseline in St. George's Respiratory Questionnaire
Description: as for outcome 6
Time Frame: Baseline, 26 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QVA149 | Tiotropium + Salmeterol/Fluticasone
Number analyzed (Participants) | 527 | 526
Score on a scale | -1.0 (0.54) | -2.5 (0.52)
Statistical Analysis 1: Comparison: QVA149 vs Tiotropium + Salmeterol/Fluticasone; Test type: Superiority; p = 0.0221, Mixed Model for Repeated measures Analys — 2-Sided; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [0.2 to 2.6]

8. Secondary Outcome: Transition Dyspnea Index (TDI) Score
Description: Transitional Dyspnea Index (TDI) score presents the degree of impairment due to dyspnea. The lower the score the worse the severity of dyspnea. The Baseline Dyspnea Index (BDI) / TDI is an instrument used to assess a participant's level of dyspnea. The BDI and TDI each have three domains: functional impairment, magnitude of task and magnitude of effort. BDI domains were rated from 0 (severe) to 4 (unimpaired) and rates summed for baseline focal score ranged from 0 to 12; lower scores mean worse severity. TDI domains were rated from -3 (major deterioration) to 3 (major improvement) and rates summed for transition focal score ranged from -9 to 9; negative scores indicate deterioration. A TDI focal score of ≥1 was defined as a clinically important improvement from baseline.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QVA149 | Tiotropium + Salmeterol/Fluticasone
Number analyzed (Participants) | 527 | 526
Score on a scale | 1.177 (0.1558) | 1.418 (0.1508)
Statistical Analysis 1: Comparison: QVA149 vs Tiotropium + Salmeterol/Fluticasone; Test type: Superiority; p = 0.1724, Mixed Model for Repeated Measures Analys; Mean Difference (Final Values) = -0.241, 95% CI [-0.587 to 0.105]

9. Secondary Outcome: Transition Dyspnea Index (TDI) Score
Description: as for outcome 8
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QVA149 | Tiotropium + Salmeterol/Fluticasone
Number analyzed (Participants) | 527 | 526
Score on a scale | 1.382 (0.1567) | 1.671 (0.1519)
Statistical Analysis 1: Comparison: QVA149 vs Tiotropium + Salmeterol/Fluticasone; Test type: Superiority; p = 0.1055, Mixed Model for Repated Measures Analysi — 2-Sided; Mean Difference (Final Values) = -0.288, 95% CI [-0.638 to 0.061]

10. Secondary Outcome: Change From Baseline in the Mean Daily Number of Puffs of Rescue Medication
Description: Change from baseline in mean daily number of puffs of rescue medication (number of puffs taken in the previous 12 hours) over 26 weeks of treatment.
Time Frame: Baseline, 26 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number of puffs per day
Arm/Group | QVA149 | Tiotropium + Salmeterol/Fluticasone
Number analyzed (Participants) | 527 | 526
Number of puffs per day | -0.307 (0.1006) | -0.484 (0.0983)
Statistical Analysis 1: Comparison: QVA149 vs Tiotropium + Salmeterol/Fluticasone; Test type: Superiority; p = 0.0641, Linear Mixed Model Analysis — 2-Sided; Mean Difference (Final Values) = 0.177, 95% CI [-0.010 to 0.365]

11. Secondary Outcome: Mean Change From Baseline in Forced Vital Capacity (FVC)
Description: Change from baseline in forced vital capacity following 26 weeks of treatment. Trough FVC is defined as the average of the pre-dose FVC measurements at -45 min and -15 min prior to dosing at each visit except Day 182 which is the average of the post-dose FVC measurements at 23h15min and 23h45min after dosing at Day 181. Baseline is considered the Day 1 average of pre-dose measurements.
Time Frame: Baseline, 26 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Tiotropium + Salmeterol/Fluticasone
Number analyzed (Participants) | 527 | 526
Liters | -0.030 (0.0192) | -0.048 (0.0186)
Statistical Analysis 1: Comparison: QVA149 vs Tiotropium + Salmeterol/Fluticasone; Test type: Superiority; p = 0.4107, Mixed Model for Repeated Measures Analys — 2-Sided; Mean Difference (Final Values) = 0.018, 95% CI 2-sided [-0.025 to 0.061]

ADVERSE EVENTS:
Time Frame: The study consists of four epochs: screening (1 week), run-in (4 weeks), blinded treatment (26 weeks) and follow-up (4 weeks).
Groups:
- Tio+Salm/Flut: tiotropium (18 μg o.d.), and salmeterol/fluticasone propionate FDC (50/500 μg b.i.d.)
Arm/Group | QVA149 | Tio+Salm/Flut
All-Cause Mortality (participants affected / at risk) | 4/527 | 5/526
Serious Adverse Events (participants affected / at risk) | 32/527 | 34/526
Other Adverse Events (participants affected / at risk) | 398/527 | 392/526
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=527) | Tio+Salm/Flut (N=526)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 3
Soft tissue infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 12 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=527) | Tio+Salm/Flut (N=526)
Atrioventricular block first degree (Cardiac disorders) | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 3 | 6
Non-cardiac chest pain (General disorders) | 3 | 6
Oedema peripheral (General disorders) | 7 | 3
Bronchitis (Infections and infestations) | 13 | 5
Influenza (Infections and infestations) | 6 | 6
Oral candidiasis (Infections and infestations) | 12 | 18
Oropharyngeal candidiasis (Infections and infestations) | 6 | 7
Pneumonia (Infections and infestations) | 2 | 6
Respiratory tract infection viral (Infections and infestations) | 1 | 6
Upper respiratory tract infection bacterial (Infections and infestations) | 2 | 6
Urinary tract infection (Infections and infestations) | 7 | 1
Viral upper respiratory tract infection (Infections and infestations) | 57 | 59
Blood creatinine increased (Investigations) | 26 | 24
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 6
Headache (Nervous system disorders) | 7 | 13
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 370 | 353
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 15
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Hypertension (Vascular disorders) | 7 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT02603393/SAP_000.pdf
  • Study Protocol (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT02603393/Prot_001.pdf